CLINICAL TRIAL: NCT03173040
Title: The Efficacy of the Traditional Chinese Medicine Niubang Pill Combined With Methotrexate on Active Rheumatoid Arthritis: a Study Protocol for a Multicenter, Randomized, Controlled Clinical Trial
Brief Title: The Efficacy of the Traditional Chinese Medicine Niubang Pill Combined With Methotrexate on Active Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cui xuejun (Other)
Collaborators: Shanghai Yueyang Integrated Medicine Hospital (Other); Longhua Hospital (Other); Shanghai 7th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Cui xuejun, Director, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Niubang Pill
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Niu Bang Zi Pill; Rheumatoid Arthritis
Keywords: Traditional Chinese medicine; Niu Bang Zi pill; methotrexate; active rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NiuBangZi pill group (Experimental): Drug: NiuBangZi pill (4g, twice a day, 3 months, oral) Drug: methotrexate (5mg, once a week, 3 months, oral) participants should administrate both NiuBangZi pill and methotrexate
  Interventions: Drug: NiuBangZi pill or NiuBangZi pill placebo
- Placeo group (Placebo Comparator): Drug: NiuBangZi placebo pill (4g, twice a day, 3 months, oral) Drug: methotrexate (5mg, once a week, 3 months, oral) participants should administrate both NiuBangZi placebo pill and methotrexate
  Interventions: Drug: NiuBangZi pill or NiuBangZi pill placebo

INTERVENTIONS:
Drug: NiuBangZi pill or NiuBangZi pill placebo — For the treatment group (NiuBangZi pill group), patients will be instructed to dissolve NiuBangZi pill (4 g) in 200 mL hot water and take the solution orally twice a day for 3 months. While patients in the placebo group will take NiuBangZi pill placebo as the same way. Besides that, both groups will also administrate MTX (5 mg per week) in addition, and glucocorticoid (less than 5mg a day) if necessary, but any other drugs especially herbs not permit.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic, systemic, inflammatory autoimmune disease that results in the destruction of joints, connective tissues, muscle, tendons and fibrous tissue. Effective therapy to manage RA still does not exit at present. Jia Wei Niu Bang Zi pill (NBZP) consists of Chinese herbals which has been widely used in the treatment of RA patients in China for hundreds of years to relieve pain and prevent the affected joints pejorative. However, there is no systematic trials to prove the effect of NBZP for management of RA.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled clinical trials will be conducted to determine whether the NBZP could make an effect of pain relief and joints protection. 120 patients suffering from active RA will be enrolled and treated with NBZP or placebo for 3 months. The primary outcome measures are the rate of American College of Rheumatology (ACR) 50, changes of the Disease Activity Score (DAS) 28 from the baseline to 3 months and the van der Heijde modified Sharp score would be measured from the baseline to 12 months. The second outcome measures are the change rate of ACR20, ACR70, Health Assessment Questionnaire - Disability Index, change score of Patient Assessment of Arthritis Pain, Patient Global Assessment of Arthritis, Patient Global Assessment of Arthritis and the Athens Insomnia Scale (AIS) from the baseline to 2 weeks, 1 month, 2 months, 3 months, 6 months, and 12 months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults with rheumatoid arthritis (score more then 5 of ACR (American College Of Rheumatology) /EULAR (European League Against Rheumatism), 2009 )
* moderate-to-severe disease activity (Disease Activity Score for 28-joint counts (DAS28) of more than 3.2
* an onset of symptoms within 12 months before enrollment, no prior exposure to more than 10mg oral glucocorticoids or biologic agents
* paid employment or unpaid but measurable work (e.g. caring for a family and home)

Exclusion Criteria:

* combined with other disease such as adjuvant arthritis, lupus arthritis, osteoarthritis and et al.
* abnormal liver and my kidney function
* pregnancy or have a plan of pregnancy,breast feeding women
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of ACR (American College of Rheumatology) 50 | at 3 months
changes of The Disease Activity Score (DAS) 28 | from baseline to 3 months
changes of the van der Heijde modified Sharp score | from baseline to 3 months

SECONDARY OUTCOMES:
changes of The Disease Activity Score (DAS) 28 | from baseline to 2 weeks
changes of The Disease Activity Score (DAS) 28 | from baseline to 1 month
changes of The Disease Activity Score (DAS) 28 | from baseline to 6 months
changes of The Disease Activity Score (DAS) 28 | from baseline to 12 months
Rate of ACR (American College of Rheumatology) 50 | at 2 weeks
Rate of ACR (American College of Rheumatology) 50 | at 1 month
Rate of ACR (American College of Rheumatology) 50 | at 2 months
Rate of ACR (American College of Rheumatology) 50 | at 6 months
Rate of ACR (American College of Rheumatology) 50 | at 12 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 weeks
change score of Health Assessment Questionnaire - Disability Index | from baseline to 1 month
change score of Health Assessment Questionnaire - Disability Index | from baseline to 2 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 3 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 6 months
change score of Health Assessment Questionnaire - Disability Index | from baseline to 12 months
change score of Patient Assessment of Arthritis Pain | from baseline to 2 weeks
change score of Patient Assessment of Arthritis Pain | from baseline to 1 month
change score of Patient Assessment of Arthritis Pain | from baseline to 2 months
change score of Patient Assessment of Arthritis Pain | from baseline to 3 months
change score of Patient Assessment of Arthritis Pain | from baseline to 6 months
change score of Patient Assessment of Arthritis Pain | from baseline to 12 months
change score of Patient Global Assessment of Arthritis | from baseline to 2 weeks
change score of Patient Global Assessment of Arthritis | from baseline to 1 month
change score of Patient Global Assessment of Arthritis | from baseline to 2 months
change score of Patient Global Assessment of Arthritis | from baseline to 3 months
change score of Patient Global Assessment of Arthritis | from baseline to 6 months
change score of Patient Global Assessment of Arthritis | from baseline to 12 months
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 2 weeks
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 1 month
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 2 months
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 3 months
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 6 months
change score of 36-item Short-Form Health Survey Questionnaire | from baseline to 12 months
change score of MOS Sleep Scale | from baseline to 2 weeks
change score of MOS Sleep Scale | from baseline to 1 month
change score of MOS Sleep Scale | from baseline to 2 months
change score of MOS Sleep Scale | from baseline to 3 months
change score of MOS Sleep Scale | from baseline to 6 months
change score of MOS Sleep Scale | from baseline to 12 months
rate of ACR20 | at 2 weeks
rate of ACR20 | at 1 month
rate of ACR20 | at 2 months
rate of ACR20 | at 3 months
rate of ACR20 | at 6 months
rate of ACR20 | at 12 months
rate of ACR70 | at 2 weeks
rate of ACR70 | at 1 month
rate of ACR70 | at 2 months
rate of ACR70 | at 3 months
rate of ACR70 | at 6 months
rate of ACR70 | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang YR, Liu L, Wang XY, Wang Q, Yao M, Cui XJ, Mao JC, Liu J, Gu XH, Chen YL, Yu X, Shi Q, Liang QQ, Wang YJ. The efficacy of the traditional Chinese medicine Jia Wei Niu Bang Zi granule combined with methotrexate in treating active rheumatoid arthritis: A multicenter, randomized, double-blinded controlled clinical trial. Medicine (Baltimore). 2019 Feb;98(6):e14424. doi: 10.1097/MD.0000000000014424. PMID 30732199